CLINICAL TRIAL: NCT05510518
Title: Late Gestational Diabetes Mellitus Diagnosis in Obese Women
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, Dr. Maya Wolf, Director of the Maternal and Fetal Medicine Unit, Western Galilee Hospital-Nahariya
Other Study IDs: 0115-22-NHR
Record Dates: First submitted 2022-07-28; First posted 2022-08-22 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy; Macrosomia, Fetal; Dystocia, Shoulder; Neonatal Jaundice; Polycythemia; Hypoglycemia Neonatal; Obesity; Obesity, Morbid
Keywords: gestational diabetes mellitus; fetal macrosomia; shoulder dystocia; maternal obesity; maternal morbid obesity
MeSH Terms: conditions — Fetal Macrosomia; Shoulder Dystocia; Jaundice, Neonatal; Polycythemia; Obesity; Obesity, Morbid; Diabetes, Gestational; Pregnancy in Obesity | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- BMI >30 kg/m2: Singleton pregnant women with normal OGTT at 24-28 weeks of gestation and BMI >30 kg/m2
  Interventions: Diagnostic Test: oral glucose tolerance test (OGTT)
- BMI >35 kg/m2: Singleton pregnant women with normal OGTT at 24-28 weeks of gestation and BMI >35 kg/m2
  Interventions: Diagnostic Test: oral glucose tolerance test (OGTT)

INTERVENTIONS:
Diagnostic Test: oral glucose tolerance test (OGTT) — • The OGTT involves assessing fasting blood glucose, drinking a solution comprising 100 g of glucose, and three glucose tests at one, two, and three hours following glucose load.

SUMMARY:
In the current work, we aim to perform a prospective study that will investigate the relationship between maternal obesity (BMI >30 kg/m2) and morbid obesity (BMI >35 kg/m2) with a late GDM diagnosis (>32 weeks), with an emphasis on obstetric and neonatal outcomes.

DETAILED DESCRIPTION:
Methods

Study design:

A prospective study that will evaluate the rate of diagnosis of late GDM and clinical effect of performing a repeat OGTT beyond week 32 in women with obesity (BMI >30 kg/m2) and morbid obesity (BMI >35 kg/m2) for whom loading sugar was normal in the second trimester. The study will be carried out in the Mother and Fetus Unit at the Galilee Medical Center in Nahariya, Israel.

Study population:

Target population: women hospitalized in the Mother and Fetus Unit for various reasons, e.g., premature labor, amniotic fluid leakage, reduced fetal movements, following a car accident, etc.

Inclusion criteria:

1. Women with normal OGTT at weeks 24-28
2. Women with BMI >30 kg/m2

Exclusion criteria:

1. Twins
2. Fetal abnormalities
3. Women who received steroids within the preceding week We will invite women who meet the enrollment criteria to participate in the study, and perform an OGTT.

Research objectives:

1. Primary endpoints:

   The percentage of obese women with late GDM diagnosis will be divided into two groups according to BMI:
   * BMI 30-35 kg/m2
   * BMI >35 kg/m2
2. Secondary endpoints:

   * Differences in the following obstetric outcomes between women diagnosed or not diagnosed with GDM: percentage of macrosomia, delivery method, shoulder dystocia, grade 3-4 tear
   * Differences in the following newborn outcomes between women diagnosed or not diagnosed with GDM: hypoglycemia, jaundice, need for phototherapy, polycythemia, hospitalization in neonatal intensive care, Apgar score, and newborn pH

Research procedure, interpretation of results, and patient follow-up:

* The OGTT involves assessing fasting blood glucose, drinking a solution comprising 100 g of glucose, and three glucose tests at one, two, and three hours following glucose load.
* Interpretation of the OGTT result is performed according to Carpenter-Coustan criteria [6]
* Women who are not diagnosed with GDM will be discharged for continued follow-up for regular prenatal care and the reason for her hospitalization.
* Per standard of care (regardless of research involvement) women diagnosed with GDM will receive counseling by a dietitian and other key department staff and undergo a complete glucose curve (seven tests per day: fasting, before each of three meals, and two hours after each meal).
* If more than 30% of glucose tests are abnormal, the patient will receive standard drug treatment.
* Follow-up is usually performed for 1-2 days in the hospital ward, after which women are discharged to ambulatory follow-up at the Mother and Fetus Clinic of the medical center.

Statistical analysis:

The sample size was calculated using the chi square formula for comparing two groups.

In a previous study in which repeat OGTT was performed beyond week 32 after initially normal results at week 24-28, the diagnosis rate of GDM for the total sample was 10%. An effect size of 20% was considered significant between obese and morbidly obese women with alpha=0.05, power 80%. The calculated sample size was 124 (at least 62 obese and 62 morbidly obese women).

ELIGIBILITY:
Inclusion Criteria:

1. Women with normal OGTT at weeks 24-28
2. Women with BMI >30 kg/m2

Exclusion Criteria:

1. Multiple pregnancy
2. Fetal defects
3. Women who received steroids within the preceding week

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women hospitalized in the Mother and Fetus Unit for various reasons, e.g., premature labor, amniotic fluid leakage, reduced fetal movements, following a car accident, etc.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Number of obese women that will be diagnosed with late GDM diagnosis by the OGTT | through study completion, an average of 1 year
  The percentage of obese women with late GDM diagnosis will be analyzed per BMI group:
  * BMI 30-35 kg/m2
  * BMI >35 kg/m2

SECONDARY OUTCOMES:
neonatal macrosomia rate | From admission to discharge, up to 1 week
neonatal hypoglycemia rate | From neonatal admission to discharge, up to 1 week
neonatal hospitalization in intensive care rate | From neonatal admission to discharge, up to 4 week

CONTACTS AND LOCATIONS:
Locations (1):
- Galil Medical Center, Nahariya, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hales CM, Carroll MD, Fryar CD, Ogden CL. Prevalence of Obesity and Severe Obesity Among Adults: United States, 2017-2018. NCHS Data Brief. 2020 Feb;(360):1-8. PMID 32487284
- [Background] Arabin B, Stupin JH. Overweight and Obesity before, during and after Pregnancy: Part 2: Evidence-based Risk Factors and Interventions. Geburtshilfe Frauenheilkd. 2014 Jul;74(7):646-655. doi: 10.1055/s-0034-1368462. PMID 25100879
- [Background] Abu Shqara R, Or S, Wiener Y, Lowenstein L, Frank Wolf M. Clinical implications of the 100-g oral glucose tolerance test in the third trimester. Arch Gynecol Obstet. 2023 Feb;307(2):421-429. doi: 10.1007/s00404-022-06520-5. Epub 2022 Mar 28. PMID 35344083
- [Background] Zilberberg E, Mazaki S, Zilberman N, Mazkereth R, Weisz B, Sivan E, et al. Should late third trimester oral glucose tolerance test be offered for patients with suspected macrosomia or polyhydramnios? Evidence in support of the clinical importance of this policy. Am J Obstet Gynecol. 2012;206(1):S122.
- [Background] Kandauda C, Wanasinghe W. Repeat OGTT at 34 - 36 weeks to detect the late occurrence of GDM: A descriptive cross-sectional study conducted at the professorial unit, teaching hospital Peradeniya, Sri Lanka. Adv Reproduct Sci. 2020;8:157-65.
- [Background] Carpenter MW, Coustan DR. Criteria for screening tests for gestational diabetes. Am J Obstet Gynecol. 1982 Dec 1;144(7):768-73. doi: 10.1016/0002-9378(82)90349-0. PMID 7148898
- [Background] Harrison RK, Cruz M, Wong A, Davitt C, Palatnik A. The timing of initiation of pharmacotherapy for women with gestational diabetes mellitus. BMC Pregnancy Childbirth. 2020 Dec 11;20(1):773. doi: 10.1186/s12884-020-03449-y. PMID 33308193